CLINICAL TRIAL: NCT03066661
Title: Expanded Access to Entrectinib (RXDX-101) for the Treatment of Cancers With NTRK, ROS1, or ALK Gene Fusions
Brief Title: Expanded Access to Entrectinib for Cancers With NTRK1/2/3, ROS1, or ALK Gene Fusions
Status: No longer available | Type: Expanded Access
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: Entrectinib (RXDX-101) - EAP
Record Dates: First submitted 2017-02-23; First posted 2017-02-28 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Cancers With NTRK, ROS1, or ALK Gene Fusions
MeSH Terms: interventions — entrectinib

INTERVENTIONS:
Drug: Entrectinib — Open-label expanded access, capsules
  Other Names: RXDX-101

SUMMARY:
Expanded access to entrectinib will be given to patients with cancers harboring NTRK1/2/3, ROS1, or ALK gene fusions who do not qualify for participation in, or who are otherwise unable to access, an ongoing clinical trial for entrectinib.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced cancer with an NTRK1, NTRK2, NTRK3, ROS1, or ALK gene fusion
* Unable to participate in an ongoing entrectinib (RXDX-101) clinical trial
* Willing and able to provide written, signed informed consent
* Medically suitable for treatment with entrectinib (RXDX-101)

Exclusion Criteria:

* Currently enrolled in an ongoing clinical study with any other investigational agent

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- 1-844-Startrk (782-7875), San Diego, California, United States